CLINICAL TRIAL: NCT02182557
Title: Phase III Double-Blind Comparative Study of WAL 801 CL Dry Syrup in Paediatric Atopic Dermatitis Patients
Brief Title: WAL 801 CL Dry Syrup in Paediatric Atopic Dermatitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 262.259
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

ARMS (2):
- WAL 801 CL Dry Syrup + Placebo (Experimental)
  Interventions: Drug: WAL 801 CL Dry Syrup; Drug: Ketotifen Fumarate Dry Syrup placebo
- Ketotifen Fumarate Dry Syrup + Placebo (Active Comparator)
  Interventions: Drug: Ketotifen Fumarate Dry Syrup; Drug: WAL 801 CL Dry Syrup placebo

INTERVENTIONS:
Drug: WAL 801 CL Dry Syrup
  Arms: WAL 801 CL Dry Syrup + Placebo
Drug: Ketotifen Fumarate Dry Syrup
  Arms: Ketotifen Fumarate Dry Syrup + Placebo
Drug: WAL 801 CL Dry Syrup placebo
  Arms: Ketotifen Fumarate Dry Syrup + Placebo
Drug: Ketotifen Fumarate Dry Syrup placebo
  Arms: WAL 801 CL Dry Syrup + Placebo

SUMMARY:
Study to investigate the safety and efficacy of WAL 801 CL Dry Syrup on pruritus associated with paediatric atopic dermatitis in comparison with that of Ketotifen Fumarate Dry Syrup and to confirm the appropriateness of dosage of WAL801 Dry Syrup.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in this study, patients must be pediatric atopic dermatitis patients that meet the following criteria and thus be appropriate for observation of pruritus. Diagnosis of atopic dermatitis was conducted in accordance with the "Definition and Diagnostic Criteria of Atopic Dermatitis" issued by the Japanese Dermatological Association.

* 15 years of age or younger
* Body weight of 14 kg or more
* Outpatients
* One week or longer has passed since the patient started to use an external steroid preparation at "Strong" or lower grade, or stopped using any external steroid preparation, at the time of obtainment of consent from the patient
* Pruritus with "2" or higher grade, immediately before initial administration

Exclusion Criteria:

* Use of sustained release adrenocorticotropic hormone (Kenacort® A, Depo-medrol®, etc.), oral preparation of methotrexate, or oral preparation of ciclosporin, within 4 weeks before initial administration of the investigational product
* Oral intake, inhalation and injection of any steroid within 2 weeks before initial administration of the investigational product
* Use of any external steroid preparation at "Very Strong" or higher grade in any sites other than the face or scalp within 2 weeks before initial administration of the investigational product
* Undergoing phototherapy
* Undergoing specific desensitization therapy or modulation therapy
* Past history of contact dermatitis caused by external steroid preparation
* Possibility of exacerbation by an external steroid preparation of infectious skin disease caused by bacteria, fungi, or virus
* Present and past history of convulsive disorder, such as epilepsy (convulsion threshold values may be lowered by the reference drug, Ketotifen Fumarate)
* Clinically significant hepatic, renal, or cardiac disease or other complications: therefore, judgement that the patient is ineligible for inclusion in this study (Please note that patients must be excluded from the study if the patients fell under Grade 2 or more, in the MHW (Ministry of health and welfare) Adverse Reaction Severity Classification Criteria.)
* Past history of allergy to any drug
* Participation in any other clinical study, or history of participation in any other clinical study within 6 months before the date when the patient gave consent to participate in this study
* Judgement by the Principal Investigator or Investigator that the patient is ineligible for inclusion in this study

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2001-06; Primary Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Degree of pruritus | at week 4

SECONDARY OUTCOMES:
Degree of pruritus | at week 2
Degree of rash | at weeks 2 and 4
Pruritus score obtained through the itching questionnaire | at weeks 2 and 4
Impression on pruritus of the patient or the parent | at week 4
Occurrence of adverse events | up to 4 weeks
Number of patients with abnormal changes from baseline in laboratory measurements (hematological tests, blood biochemical tests, and urinalysis) | Baseline and week 4